CLINICAL TRIAL: NCT01965717
Title: Multicentre Trial Of Serum Levels Of MMP-9 As A Biomarker Of Endoleak
Acronym: BIOLEAK
Status: Completed | Type: Observational
Sponsor: Igor Koncar (Other)
Collaborators: University of Genua, Italy (Other); Charles University, Czech Republic (Other)
Responsible Party: Sponsor-Investigator, Igor Koncar, vascular surgeon, University of Belgrade
Organization: University of Belgrade (Other)
Other Study IDs: KVEH KCS
Record Dates: First submitted 2013-10-15; First posted 2013-10-18 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Endoleak After Endovascular Aneurysm Repair
Keywords: endoleak; MMP- 9; biomarker
MeSH Terms: conditions — Endoleak

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood will be drawn via an antecubital vein puncture and collected in Heparin buffered vacutainer for plasma. Exactly 30 min after collection, blood will be centrifuged (15 min, 1000 g, 4C) and multiple aliquots will be stored at exactly 1 h after collection at < - 20 C.
Oversight: Data Monitoring Committee: No

SUMMARY:
Endovascular procedures already brought enormous revolution in the process of treatment of patient with abdominal aortic aneurysm (AAA). It is well defined that early mortality and morbidity is significantly reduced comparing to open repair. The persistent concern is long term durability of devices and their success of aneurysm exclusion in order to prevent rupture. At the moment the best armament to prevent rupture after endovascular exclusion is the watchful waiting and timely reintervention. The main complication that follows this procedure and causing catastrophic long term complications is endoleak. The ideal algorithm to follow up patients after aneurysm exclusion has not been found. In order to reveal endoleak ultrasound is used more than before, however frequent computerized tomography is wasting a lot of costs and exposing patients to irradiation and nephrotoxic contrast.

Matrix metalloproteinase activity has been demonstrated in the process of aneurysm development. Imbalance between MMP and its inhibitors TIMP provokes collagenolytic and elastolytic activity that is inducing aneurysmatic degeneration of aortic wall. Due to the previously described connection between aneurysm and MMP activity, it was proved that serum level of MMP-9 is significantly higher in patients with abdominal aortic aneurysm (AAA). Also, higher levels of MMP-9 were discovered in patients with inadequate aneurysm exclusion after endovascular procedure suggesting that degradation of the aortic wall is still ongoing process, not being the case with successfully excluded aneurysm. There might be a potential role of MMP-9 serum level as a biomarker of present endoleak after endovascular aneurysm exclusion.

All published trials have shown correlation between MMP 9 activity and presence of endoleak, however, no correlation was made between specific types of endoleak and necessity to reoperation (clinical significance). Additionally there were only four trials presented in the literature investigating low number of patients.

Since there is possible value of MMP-9 serum level as biomarker of present endoleak, further studies are necessary. This why we are organizing multicentre trial, that will cover significant number of patients in order to define

* Value of MMP-9 as a biomarker of successful initial exclusion
* Value of MMP-9 level as predictor of aneurysm shrinkage
* Value of MMP-9 level in patients with increased aneurysm diameter and no visible endoleak
* Correlation of the MMP -9 serum level with different type of enoleak
* Value of MMP-9 as biomarker of successful treatment of endoelak

Material and methods Patient with AAA greater then 55 mm in diameter that are candidates for endovascular repair will be selected. Demographic, anatomical and data regarding the procedure will be gathered prospectively. Also serum levels of MMP-9 will be measured before procedure, during the first week before discharge, and after 1,6,12,18,24,36,48 months. On the same day of measuring MMP-9 level control MSCT and ultrasonography exam will be performed in order to collect data regarding the success of exclusion and presence of any endoleak with the accurate measurement of aneurysm diameter changes. Ultrasonography and MSCT exam will be performed by experienced physicians, also preoperative evaluation of anatomical data.

In case of reintervention additional questionnaire will be filled regarding anatomical and procedure related data using pre and postoperative ultrasound and MSCT examination, while MMP-9 levels will be measured before procedure and after the procedure using the same protocol as for primary procedure.

Statistical analysys Levels of MMP-9 in serum with presence of different types of endoleak will be correlated one week and 1,6,12,18,24,36 48 months after the procedure Anatomical data will be correlated with the decrease in MMP-9 level before and after procedure Levels of MMP-9 in serum after one week and one month will be correlated with further aneurysm shrinkage Level of MMP-9 in serum with type of endoleak will be correlated Level of MMP-9 before and after reoperation will be compared Level of MMp-9 in serum of patients with disappearing endoleaks will be followed Level of MMP-9 in serum of patients with new endoleaks will be followed

DETAILED DESCRIPTION:
1. Summary

   Endovascular aortic aneurysm repair (EVAR) provides low early mortality and requires intensive follow up of the patients in order to prevent rupture as a consequence of endoleak. Follow up protocols are changing with time differing between the hospitals and even the physicians. Ultrasonography (US), contrast enhanced ultrasonography, multisliced computed tomography (MSCT) and native radiography are most frequently used. All these techniques are combined in order to compensate their lacks and disadvantages. The new methods for early detection of endoleak should improve this cumbersome follow up process.

   Matrix metalloproteinase (MMP) activity has been demonstrated in the process of aneurysm development. Higher level of MMP-9 were discovered in patients with inadequate aneurysm exclusion after endovascular procedure suggests that degradation of the aortic wall is still ongoing process and that there might be a potential role of MMP-9 serum level as a biomarker in endoleak detection.

   Aim of this study is to explore the serum levels of MMP - 9 in patients treated with endovascular aneurysm repair and to provide some more profound information regarding its' correlation with different types of endoleak.

   Patients treated with EVAR will be followed for at least one year. During five visits, with first preoperative, then on discharge, and after one, six and twelve months, patients will be examined by means of US and MSCT. During the same five visits serum levels of MMP -9 will be measured and correlated with different levels of aneurysm exclusion. Collected anatomical, demographic data of the patients and intraoperative data related to the technical success of the procedure will provide subgroup of patients with higher correlation between the aneurysm exclusion and serum level of MMP -9. The primary outcome measure is the serum levels of the MMP - 9 at one, six and twelve months after treatment and its relation with anatomical, demographic and procedure related data. Clinical outcome events include different types of endoleak. The secondary outcome is the correlation of different types of endoleak with the serum levels of the MMP - 9.

   This study is designed to be multicentre and to recruit 150 patients over a 24-month period. Leading center is Clinic for Vascular and Endovascular Surgery of the Serbian Clinical centre. Participating center should be able to perform EVAR, follow up patient with US and MSCT for four times in the first year and to detect serum levels of MMP - 9. All analysis will be performed individually by participating centre encouraged to use same techniques as the leading center. Individual experience of collaborators in the participating centre will be recorded before their inclusion in the study.
2. Background

   Endovascular procedures already brought enormous revolution in the process of treatment of patient with abdominal aortic aneurysm (AAA). It is well defined that early mortality and morbidity is significantly reduced comparing to open repair. The persistent concern is long term durability of devices and their success of aneurysm exclusion in order to prevent rupture. At the moment the best armament to prevent rupture after endovascular exclusion is the watchful waiting and timely reintervention. The main complication that follows this procedure and causing catastrophic long term complications is endoleak. The ideal algorithm to follow up patients after aneurysm exclusion has not been found. In order to reveal endoleak ultrasound is used more than before, however frequent computerized tomography is wasting a lot of costs and exposing patients to irradiation and nephrotoxic contrast.

   Matrix metalloproteinase activity has been demonstrated in the process of aneurysm development. Imbalance between MMP and its inhibitors TIMP provokes colagenolitic and elastolytic activity that is inducing aneurysmatic degeneration of aortic wall. Due to the previously described connection between aneurysm and MMP activity, it was proved that serum level of MMP-9 is significantly higher in patients with abdominal aortic aneurysm (AAA). Also, higher levels of MMP-9 were discovered in patients with inadequate aneurysm exclusion after endovascular procedure suggesting that degradation of the aortic wall is still ongoing process, not being the case with successfully excluded aneurysm. There might be a potential role of MMP-9 serum level as a biomarker of present endoleak after endovascular aneurysm exclusion.

   All published trials have shown correlation between MMP 9 activity and presence of endoleak, however, no correlation was made between base levels and specific types of endoleak and necessity to reoperation (clinical significance). Additionally there were only four trials presented in the literature investigating low number of patients 1,2,3,4.
3. Aims of the trial and hypothesis

The basic research question is whether the level of MMP -9 is changing after endovascular aneurysm exclusion and what is the curve of the level of active MMP-9 concentration in the first year after the procedure. We hypothesize that the level of MMP-9 active concentration should decline, however it might be dependent on some other factors.

Secondary research questions are:

1. What is the role of pre-treatment serum levels of the MMP - 9 in patient with AAA? We hypothesized that pre operative serum levels of the MMP - 9 should be predictor of its sensitivity in endoleak detection in the postoperative follow up.
2. What is the role of the serum levels of the MMP - 9 as a biomarker of the early successful aneurysm exclusion? We hypothesize that the serum levels of the MMP - 9 in the early postoperative time (first week and one month) could be biomarker of successful aneurysm exclusion
3. What is the role of the serum levels of the MMP - 9 in differentiating the types of endoleak? We hypothesized that different serum levels of the MMP - 9 could be found in patients with different types of endoleak.
4. What is the role of the serum levels of the MMP - 9 after reintervetion due to a present endoleak? We hypothesized that the levels of endoleak should decline after successful re-treatment
5. What is the role of the serum levels of the MMP - 9 as a predictor of aneurysm sac enlargement? We hypothesized that the serum levels of the MMP - 9 in the early postoperative time (up to one month) could correlate with sac enlargement in patient with no visible endoleak .

4. Study design 4.1. Patient enrollment and data collection The BIOLEAK study is designed to become multicentre study. The minimum requirement for participation of a center in this study is to perform EVAR procedures, and to have laboratory capable of the serum levels of the MMP - 9 analyses. Center agreeing to collaborate should follow up patients with MSCT and ultrasound for minimally four times in the first year and then at least once yearly thereafter. In the same time with these follow up exams serum levels of the MMP - 9 should be measured. The preferable method of the measurement is given below; however, every center is encouraged to participate in the trial by using its own available method with previous notification and confirmation by the leading center.

All study participants will undergo 5 ultrasound and 5 MSCT exams in the first year of participation. Both MSCT and ultrasound should be performed before procedure, before discharge after the procedure, one, six and twelve months after the procedure. All preoperative anatomical and postoperative control images and ultrasound assessment should be performed by the most experienced stuff of the collaborating center. Ultrasound assessment should be made by Color duplex technique, widely used. MSCT image assessment should be made using the post processing techniques and center line analysis. Control MSCT exams should be made according to the protocol of the participating center.

Blood samples to determine serum levels of the MMP - 9 as a biomarker of the aneurysm exclusion should be obtained at five time points in the first year and analyzed individually in the laboratory of the participating center: 1- 3 days before treatment, 2-7 days after treatment, one, six and twelve months after treatment. Blood sample should be taken on the same day when performing ultrasound and/or MSCT exam. Minimum requirements for participating in the trial is to measure serum levels of the MMP - 9, however participating centre could also include in the analysis: matrix-metalloproteinases and inhibitors (MMP-1,2,3,7,10, TIMP-1). The analyzed method should be according to the capabilities of the participating centre, while the leading center Clinic for Vascular and Endovascular Surgery of the Serbian Clinical Centre will be measured serum MMP-9 levels with Fluorokine E (Human Active MMP-9 Fluorescent Assay). The process of material collection and storage was suggested by producer (R&D Systems).

Venous blood will be drawn via an antecubital vein puncture and collected in Heparin buffered vacutainer for plasma. Exactly 30 min after collection, blood will be centrifuged (15 min, 1000 g, 4C) and multiple aliquots will be stored at exactly 1 h after collection at < - 20 C.

One sample more from every visit should be stored for at least 12 months for additional analysis if necessary.

Preoperative, discharge and one month follow up samples of each patient will be measured at the same time identically in order to have same calibration and reagent.

For the collaborating centers: Usage of the same process of collecting and storing samples as well as calculating the results will contribute to the quality of results. However, this is optional condition for participating in the study and all the centers should used their own methods while the leading center should be informed about the differences in this process.

4.2. Detailed description of the data collection

Patient with inclusion criteria will be selected and after signing consent form will be included in the trial. Treating physician will report selected patient by filling the inclusion form and demographic data form and sending it to the leading center.

INCLUSION FORM should be filled and sent to the trial center together with DEMOGRAPHIC DATA FORM via fax (+381113065177). This form will include basic anatomical information regarding the patient anatomy related to the success of the procedure. All data related to the anatomical features of the treated aneurysm should be assessed by operating surgeon or radiologists, or experienced member of the team, by using center line analysis software. Extension of the aneurysm process should be defined according to the planned LZ location in the iliac zone. Collateral vessels that are patent and greater than 1 mm in diameter should be counted using the imaging detailed analysis. We are assuming that the number of collateral vessels could influence the levels of MMP -9 in the postoperative and follow up time. Surely the number of these vessels could influence the rate of endoelak type II. When filling the form "inferior mesenteric artery" should be round off or marked with "X", while the number of patent lumbal, hypogastric or accessory renal arteries that are going to be excluded should be stated in the blank line. Neck diameter should be measured in the inner to inner fashion, while in case of non cylindrical neck the greatest value should be stated. Aneurysm length should be measured from the lower renal artery to the distal end of the LZ, for the both, left and right side. Neck length is defined only as a length of the fixation zone and not the whole neck, which in case of long conical necks might be different. Neck configuration should be assessed by center line analysis and one of the offered configurations should be chosen. It is important to differ cylindrical from non cylindrical necks. Neck angulations with suprarenal aorta and aneurysm sack should be measured separately. Parietal thrombus and calcification should be expressed in percentage of the circumference and the greatest thickness diameter should be stated. Greatest aneurysm diameter, narrowest aortic lumen and lumen of the aorta at the level of bifurcation should be expressed in mm. Common iliac artery diameters should be measured in three levels, the initial, middle and the distal part at the level of iliac bifurcation, and should be expressed in mm. Iliac angulations should be measured between the aneurysm and proximal iliac center line. Name hospital and email of the corresponding physician should be stated at the end of the INCLUSION FORM.

DEMOGRAPHIC DATA FORM should be sent together with INCLUSION FORM. The presence of co-morbid conditions should be noted in this form, together with age, sex, previous surgical procedures and active medical therapy.

After sending these forms, patient will be included in the study on the intention to treat basis and corresponding physician will be informed about the PATIENT INCLUSION NUMBER. The procedure should be planned the sooner the better.

PROCEDURE FORM should be filled to a certain extent after the procedure and the second part on the discharge day. Date of the procedure and patient inclusion number should be stated. Inclusion number will already sent by email from the trial center (Clinic for Vascular and Endovascular Surgery, Serbian Clinical Center). Name of the operating surgeon and his assistant should be stated. The configuration of the stent graft chosen and implanted should be stated in the named rows (proximal stent graft diameter, distal stent graft diameter). Number of used extensions should not count body and contralateral limb as a necessary minimum, while aorto-uni configuration should be confirmed with "yer" or "no". All additional procedures performed in order to reduce the endoleak rate should be marked. If any additional are performed it should be stated in the column left for comments. Intraoperative control angio after performing total procedure should be made as common in the collaborating center, and the result should be assessed by operating surgeon. If there is uncertainty with endoleak type II it should be marked as probably. If operating surgeon is certain, it should be marked as obvious. Other measures to reduce the endoleak probability after performing control angio should be marked. The result of the angio after additional measures is not supposed to be included in the procedure form, however if there are any comments they should be stated in the column left for comments. On the discharge day all intrahospital postoperative anticoagulant therapy should be noted, complications, outcome, additional procedures and length of hospital stay.

FOLLOW UP FORM is designed to have data related to ultrasonogrpahy, MSCT follow up exams and serum levels of MMP -9 at the all five planned visits in one place. However, since the process of calculating serum levels of MMP-9 usually requires storing and gathering samples until complete kit box can be used, it may cause delay in follow up completion. Additionally results of the one month follow up will be objective of the interim analysis. For these purposes, it is necessary to send this form via fax two times. First time is after completing results for the preoperative, on discharge and one month follow up serum levels of MMP - 9 with ultrasound and MSCT analysis. Second time is when complete data for the one year follow up are collected. During all this time this form and all others should be kept with all other forms in the patients official medical documents.

4.3. Flow chart

Five study visits will be done in each patient in the first participating year as showed in the following flow-chart.

MMP9 ULTRASONOGRAPHY MSCT PREOPERATIVE X X X ON DISCHARGE (2-7 days) X X X ONE MONTH X X X SIX MONTHS X X X ONE YEAR X X X For the purposes of central data collection, all four data forms should be sent via fax to the Clinical for Vascular and Endovascular Surgery, of the Serbian Clinical Centre, +381 11 30565177.

4.4. Outcome measures The primary outcome measure is the serum levels of the MMP - 9 at one, six and twelve months after treatment and its relation with anatomical, demographic and procedure related data. Clinical outcome events include different types of endoleak. The secondary outcome is the correlation of different types of endoleak with the serum levels of the MMP - 9.

5. Safety aspects

The present study is a purely observational study and is not associated with any clinical risk for complications after edovascuar aneurysm repair. About 30 ml of blood in total will be drawn for serum analysis during all five visits in the first year. Ultrasound and MSCT imaging methods are non-invasive techniques that are part of regular follow up after endovascular aneurysm repair.

6. Statistical Analysis and sample size

6.1. Sample size justification and statistical methods The present study aims to enroll 150 patients from different high-volume centers over a recruitment period of 2 years. The serum levels of the MMP - 9 will be compared between patients and between the different visits using logistic regression models. Interactions between MMP - 9 levels and different types of endoleak will be investigated in subgroup analyses. Also interaction between anatomical data, demographic and procedural data with serum levels of the MMP - 9 , aneurysm sac size and presence of endoleak will be analyzed.

6.2. Interim analysis An interim analysis will be performed after completing one month follow up of first 30 patients in order to check the serum levels of the MMP - 9 and its calculation difficulties - if any.

7. Ethical considerations

Ultrasound and MSCT examinations detailed in the protocol are part of the routine clinical work-up in patients before and after EVAR without any known side effects in patients without contraindications. With the exception of blood sampling, no invasive examinations are made. Identifying the benefit of the serum levels of the MMP - 9 as a biomarker of endoleak could contribute to better detection of endoleak and reduce costs and efficacy of the follow up. It will support selection of different follow up protocols on the individual basis for every patient.

Participation in the BIOLEAK study is completely voluntary. Eligible patients are informed about the study by investigators and will be given written patient information. Patients willing to participate are required to provide written informed consent to participate. Study participants retain the right to withdraw their consent to participate at any time after initial consent was given, without any consequences for clinical management and standard of care received. If a patient withdraws consent or not willing to participate during the process of follow up (rejecting blood sampling or repetitive MSCT or ultrasound exam), available data should be used in the overall analysis.

8. Study management 8.1. Study management and participating centers This study is led by the Clinic for Vascular and Endovascular Surgery of the Serbian Clinical Center (lead investigator Prof Dr Lazar Davidovic). Its Serbian phase is a part of the scientific research project (No 175008) supported by the Ministry of Education and Science of the Republic of Serbia. Collaborating centres are in the process of entering the study at the moment.

All centers performing endovascular exclusion of the infrarenal abdominal aortic aneurysms with available imaging, ultrasonographic and laboratory facilities are invited to join this trial. Physicians that enroll patients into the BIOLEAK study will act as co-investigators and participate as authors in resulting publications. Center willing to participate will apply by filling the COLLABORATING CENTRE TRACK RECORD and sending it to the leading investigator - Prof Dr Lazar Davidovic at davidovic.lazar@gmail.com . In this form it is possible and encouraging to state multiple operators, ultrasonographers and MSCT reading physicians.

This is an investigator-initiated trial. The lead investigator and co-investigators will have unrestricted access to the data. The local investigators at the participating centers will meet with the lead investigator and co-investigators on a regular basis to discuss progress of recruitment and assess the quality of the acquired data. The lead investigator, co-investigators, the local ethics committee or any other supervisory body may audit or inspect the local study sites at any time. Data steering committee will be formed once this study becomes a multicentre.

8.2. Data storage and protection Documentation of the data of every study participant will be done by completing electronic forms and sent via fax to the BIOLEAK study center at the Clinic for Vascular and Endovascular Surgery of the Serbian Clinical Center. Blood samples will be separately analyzed in every participating center where will be stored and kept under the local regulations. If consent is withdrawn at any time after study entry, any blood samples obtained from the patient should be destroyed. Any results obtained from the analysis of those samples before consent was withdrawn may be used for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* Patient fulfilling criteria for endovascular repair of infrarenal abdominal aortic aneurysm according to criteria of the participating centre.

Exclusion Criteria:

* Already performed endovascular aneurysm exclusion with unknown baseline levels of MMP-9; presence of aneurysm in other location; usage of MMP-9 inhibiting drugs (tetraciklincs); presence of active malignant disease;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with implantation of endovascular stent graft due to abdominal aortic aneurysm
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2012-07; Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Level of MMP 9 | 12 months
  The primary outcome measure is the serum levels of the MMP - 9 at twelve months after treatment

SECONDARY OUTCOMES:
Correlation of presence of endoleak and level of MMP 9 | 12 months
  The secondary outcome measure is the correlation between the serum levels of the MMP - 9 at twelve months after treatment and presence of endoleak

CONTACTS AND LOCATIONS:
Overall Officials: Lazar Davidovic, Prof, Principal Investigator — Clinic for Vascular and Endovascular Surgery, Serbian Clinical Centre
Locations (1):
- Clinic for Vascular and Endovascular Surgery, Serbian Clinical Centre, Belgrade, Serbia

REFERENCES:
- [Background] Monaco M, Stassano P, Di Tommaso L, Iannelli G. Response of plasma matrix metalloproteinases and tissue inhibitor of metalloproteinases to stent-graft surgery for descending thoracic aortic aneurysms. J Thorac Cardiovasc Surg. 2007 Oct;134(4):925-31. doi: 10.1016/j.jtcvs.2007.05.044. PMID 17903509
- [Background] Lorelli DR, Jean-Claude JM, Fox CJ, Clyne J, Cambria RA, Seabrook GR, Towne JB. Response of plasma matrix metalloproteinase-9 to conventional abdominal aortic aneurysm repair or endovascular exclusion: implications for endoleak. J Vasc Surg. 2002 May;35(5):916-22. doi: 10.1067/mva.2002.123676. PMID 12021707
- [Background] Sangiorgi G, D'Averio R, Mauriello A, Bondio M, Pontillo M, Castelvecchio S, Trimarchi S, Tolva V, Nano G, Rampoldi V, Spagnoli LG, Inglese L. Plasma levels of metalloproteinases-3 and -9 as markers of successful abdominal aortic aneurysm exclusion after endovascular graft treatment. Circulation. 2001 Sep 18;104(12 Suppl 1):I288-95. doi: 10.1161/hc37t1.094596. PMID 11568071
- [Result] Hellenthal FA, Ten Bosch JA, Pulinx B, Wodzig WK, de Haan MW, Prins MH, Welten RJ, Teijink JA, Schurink GW. Plasma levels of matrix metalloproteinase-9: a possible diagnostic marker of successful endovascular aneurysm repair. Eur J Vasc Endovasc Surg. 2012 Feb;43(2):171-2. doi: 10.1016/j.ejvs.2011.10.014. Epub 2011 Dec 14. PMID 22172237